CLINICAL TRIAL: NCT06369155
Title: A Biomarker Study of the Wee1 Inhibitor Azenosertib (ZN-c3) in Women With Recurrent or Persistent Uterine Serous Carcinoma
Brief Title: Azenosertib in Uterine Serous Carcinoma: Biomarker Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joyce Liu, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Zentalis (Unknown)
Responsible Party: Sponsor-Investigator, Joyce Liu, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-061
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Uterine Serous Carcinoma; Uterine Carcinoma; Uterine Cancer
Keywords: Uterine Serous Carcinoma; Uterine Carcinoma; Uterine Cancer; Persistent Uterine Serous Carcinoma
MeSH Terms: conditions — Uterine Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azenosertib (Experimental): 25 participants will be enrolled and will complete study procedures as follows:
  * Baseline visit with assessments and CT or MRI scan.
  * CT or MRIs scans every 2 cycles.
  * Cycle 1 through End of Treatment:
    --Days 1 through 5, 8 through 12, and 15 through 19: Predetermined dose of Azenosertib 1x daily.
  * End of Treatment visit.
  Interventions: Drug: Azenosertib

INTERVENTIONS:
Drug: Azenosertib — Wee1 inhibitor, 25mg and 100mg tablets, taken orally per protocol.
  Other Names: Zn-c3; C29H34N8O2

SUMMARY:
This research study is being done to investigate how Azenosertib affects tumor cells of persistent or recurrent uterine serous carcinoma.

The name of the study drug involved in this study is:

-Azenosertib (a type of Wee1 inhibitor)

DETAILED DESCRIPTION:
This research study is being done to investigate how Azenosertib affects tumor cells of persistent or recurrent uterine serous carcinoma. Azenosertib has been tested as a treatment for other diseases and has shown to stop cancer cell growth.

The U.S. Food and Drug Administration (FDA) has not approved Azenosertib as a treatment for recurrent uterine serous carcinoma.

This research study involves screening for eligibility, study treatment visits, X-rays, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, Positron Emission Tomography CT (PET-CT) scans, Meta-iodobenzylguanidine (MIBG) scans, Fluorodeoxyglucose Positron Emission Tomography), (FDG-PET) scans, Electrocardiograms (EKGs), tumor biopsies, and blood tests.

It is expected that about 25 people will take part in this research study.

Zentalis Pharmaceuticals is supporting this research study by providing the study drug Azenosertib.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed recurrent or persistent uterine serous carcinoma. For the purposes of this study, uterine carcinomas (with the exception of carcinosarcomas) that have any component that is considered serous will be considered a uterine serous carcinoma.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured per RECIST 1.1 criteria. See Section 12 for the evaluation of measurable disease.
* Participants must have had one prior platinum-based chemotherapy regimen for management of advanced or metastatic uterine serous carcinoma. Participants with early stage disease who received adjuvant platinum-based chemotherapy are also eligible if they recur within 12 months of their adjuvant therapy. Chemotherapy administered only in conjunction with primary RT as a radiosensitizer should not count as a systemic regimen. There is no restriction on the number of prior lines of therapy a participant may have previously received. Additionally, participants must have a known tumor MSI or MMR status and those participants with MSI-high or MMR-deficient tumors must have already received prior therapy with a PD1 or PD-L1 immune checkpoint inhibitor or be deemed not to be a candidate for immune checkpoint therapy.
* Age 18 years or older. Because no dosing or adverse event data are currently available on the use of azenosertib in participants <18 years of age, children are excluded from this study.
* ECOG performance status 0, 1, or 2 (see Appendix A)
* Participants must meet the following organ and marrow function as defined below:

  * absolute neutrophil count ≥1500/mcL
  * hemoglobin ≥9 g/dL (must be at least 2 weeks since any blood transfusion)
  * platelets ≥100,000/mcL
  * total bilirubin ≤ institutional upper limit of normal (ULN) or

    ≤1.5x ULN in patients with liver metastases or well-documented Gilbert's Syndrome
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN or ≤5 × institutional ULN in patients with liver metastases
  * creatinine ≤ 1.5x institutional ULN or estimated CrCl≥ 60 mL/min
* Willingness to release archival tissue for research purposes.
* Biopsiable disease in a lesion that is not being utilized as the target lesion for RECIST assessment and willing to undergo pre- and on-treatment biopsies.
* HIV-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. However, participants who are on antiretroviral therapy that includes strong inhibitors or inducers of CYP3A4 are not eligible, given the potential for interaction with azenosertib, which is a CYP3A4 substrate.
* Participants with treated brain metastases are eligible if follow-up brain imaging after CNS-directed therapy shows no evidence of progression. Participants with new or progressive brain metastases (active brain metastases) are eligible only if the treating physician determines that immediate CNS-specific treatment is not required and is unlikely to be required during the first two cycles of therapy. Participants with known leptomeningeal disease are not eligible.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* The effects of azenosertib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy, radiotherapy, or investigational therapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to first dose of azenosertib. Participants may not have had hormonal therapy within 2 weeks of the first dose of azenosertib.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy administered more than 3 weeks before first dose of azenosertib (e.g.,., have residual toxicities > Grade 1) with the exception of alopecia.
* Participants who are receiving any other investigational agents for this condition.
* Participants may not have had prior receipt of a cell cycle checkpoint inhibitor (e.g., Chek1, Wee1, or ATR inhibition)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to azenosertib.
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine.
* Pregnant women are excluded from this study because azenosertib is an DNA damage repair pathway agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with azenosertib, breastfeeding should be discontinued if the mother is treated with azenosertib.

  --Women of childbearing potential (WoCBP) may be included only if acceptable contraception (see Appendix C) is in place for two weeks before study entry, for the duration of the treatment with the study drug and for 5x half-lives of ZN-c3 + 6 months after the last dose of ZN-c3. Sexually active female subjects of childbearing potential must agree to use protocol-recommended method of contraception from the start of the screening period until 6 months after the last dose of study drug ZN-c3.
* Participants must not have undergone major surgical procedures within 28 days of beginning study treatment or minor surgical procedures within 7 days of beginning study treatment. Port-a-cath placement will be allowed within a 7 day window of starting study treatment.
* Participants must be able to swallow oral medication and may not have refractory nausea and vomiting, have a percutaneous endoscopic gastrostomy (PEG) tube, be receiving total parenteral nutrition (TPN), or be dependent on IV fluid support.
* Because the composition, PK, and metabolism of many herbal supplements are unknown, the concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, cannabis, St. John's wort, kava, ephedra [ma huang], ginkgo biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, and ginseng). Participants should stop herbal medications at least 7 days prior to first dose of azenosertib.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in Replication Fork Speed in Overall Response | Up to 7 months
  Replication fork speed assessed by DNA fiber assays in PDO models. Responder defined as participants achieving complete response (CR) or partial response (PR) based on RECISTv1.1 criteria. Wilcoxon rank sum tests will be used to compare the percentage change in replication fork speed with exposure to WEE1 inhibition in co-clinical models between overall response responder and non-responder.
Percentage Change in Replication Fork Speed in 6 Month Progression Free Survival (PFS6) | At 6 months
  Replication fork speed assessed by DNA fiber assays in PDO models. PFS6 is a binary endpoint where patients that are alive and progression free (per RECIST 1.1) at 6 months are considered responders. All other patients (those that died or progressed prior to 6 months or those with less than 6 months of follow-up for progression) are considered non-responders. Wilcoxon rank sum tests will be used to compare the percentage change in replication fork speed with exposure to WEE1 inhibition in co-clinical models between overall response responder and non-responder.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 7 months
  The overall response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECISTv1.1 criteria.
6-month Progression-Free Survival (PFS6) | At 6 months
  6-month PFS is a probability estimated using progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) or death, or is censored at time of last disease assessment.
Clinical Benefit Rate (CBR) | Up to 7 months
  CBR defined as proportion of participants with Partial Response (PR) + Complete Response (CR) + Stable Disease (SD) ≥6 months per RECIST 1.1
Median Duration of Overall Response (DOR) | Up to 7 months
  Duration of Overall Response (DOR), estimated using the Kaplan Meier method, is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) per RECISTv1.1, until the first date that recurrent or progressive disease is objectively documented. Participants without progressive disease are censored at the date of last disease assessment.
Median Progression-Free Survival (PFS) | 2 years
  Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) or death, or is censored at time of last disease assessment.
Grade 3-5 Treatment-related Toxicity Rate | Up to 7 months
  All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 that are not resolved in accordance with treatment guidelines were counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Liu, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu